CLINICAL TRIAL: NCT05448001
Title: A Multi-center, Randomized, Double-Blind, Active-Controlled, Parallel Group, Phase III Clinical Trial to Evaluate the Efficacy and Safety of JP-1366 in Patients With Gastric Ulcer
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of JP-1366 in Patients With Gastric Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP-1366-303
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Gastric Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental)
  Interventions: Drug: JP-1366 20mg
- Control Group (Active Comparator)
  Interventions: Drug: Lansoprazole 30mg

INTERVENTIONS:
Drug: JP-1366 20mg — JP-1366 20 mg 1 capsule, Lansoprazole 30 mg placebo 1 capsule before meal
  Arms: Study Group
Drug: Lansoprazole 30mg — JP-1366 20 mg placebo 1 capsule, Lansoprazole 30 mg 1 capsule before meal
  Arms: Control Group

SUMMARY:
A Multi-center, Randomized, Double-Blind, Active-Controlled, Parallel Group, Phase III Clinical Trial to Evaluate the Efficacy and Safety of JP-1366 in Patients with Gastric Ulcer

ELIGIBILITY:
* Inclusion Criteria: Subjects who meet all of the following criteria can participate in this study:

  1. Male or female, ≥ 19 years of age at the time of obtaining consent
  2. Confirmation via upper gastrointestinal endoscopy within 14 days from Visit 2 for the following:

     º One or more GUs with the largest ulcer ≥ 3 mm to ≤ 30 mm

     º Largest ulcer classified as A1 or A2 based on Sakita-Miwa classification
  3. Subjects who fully understand this study and voluntarily signed the informed consent form
* Exclusion Criteria: Subjects who meet any of the following criteria cannot participate in this trial:

[Medical History]

1. Subjects who have undergone gastric acid secretion suppression surgery, gastric surgery (e.g., gastrectomy and gastromucosectomy), resection of entire small bowel (excluding simple ulcer closure and endoscopic benign tumor resection) or esophageal surgery
2. Subjects with history of Zollinger-Ellison syndrome or gastric hypersecretion
3. Subjects with hypersensitivity (present or past) to any substance in the IP, drugs in the same class as them (potassium-competitive acid blocker [P-CAB] and proton pump ingibitor[PPI]), or benzimidazole
4. Subjects with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
5. Subjects with malignant gastrointestinal cancer regardless of the period, Subjects with a history of malignancy within 5 years from Visit 1 (however, subjects with basal cell carcinoma or squamous cell carcinoma who require steady long-term follow-up only without therapeutic dosing/procedure/surgery, etc. can participate in this trial)
6. Subjects with a history of drug or alcohol abuse within 1 year from Visit 1.
7. Subjects who have had or are scheduled to have major surgery that may affect gastric acid secretion within 30 days from Visit 1

   [Comorbidity]
8. Subjects with gastrointestinal bleeding, esophageal stricture, ulcer-induced stenosis, pyloric stenosis, gastroesophageal varices, Barrett's esophagus (> 3 cm), esophageal dysplasia, duodenal ulcer, glandular ulcer, refractory ulcer, perforation ulcer, or surgery-induced ulcer at Visit 1
9. Subjects with signal symptoms (dysphagia, severe dysphagia, bleeding, weight loss, anemia, and bloody stools) that suggest malignant tumors of gastrointestinal tract at Visit 1 (except a tumor confirmed negative in endoscopy, etc.)
10. Subjects with pancreatitis, inflammatory bowel Disease (Crohn's disease, ulcerative colitis, or Behcet's enteritis) at Visit 1
11. Subjects with known acquired immune deficiency syndrome (AIDS) or hepatitis (including Hepatitis B surface (HBs) antigen positive, Hepatitis C virus (HCV) antibody positive, or hepatitis virus carrier) (except subjects that are HCV-RNA negative)
12. Subject with clinically significant mental illness
13. Thrombotic patients (cerebral thrombosis, myocardial infarction, thrombophlebitis, etc.)
14. Subjects who confirmed malignant tumors by upper gastrointestinal endoscopy during the Screening (Visit 1). If a biopsy is required. Subject who may have an impact on the lesion evaluated in this clinical trial needs to be excluded, and the biopsy should not be delayed for registration in this clinical trial.

    [Drug Dosing/Treatment History]
15. Subjects with a history of taking any of the following drugs or those required to take them until the end of treatment (EOT): For participation in this trial, stable drugs must not be discontinued.:

    <Drugs prohibited from within 2 weeks of Visit 1 to EOT>

    º All acid blockers other than the IPs: H2 receptor antagonists, proton pump inhibitors (PPIs) and potassium-competitive gastric acid blockers

    º Gastromucosal protection agents: Prostaglandins (however, local administration is allowed) and mucosal blood flow stimulants Antacids

    º Gastrointestinal motility stimulants

    º Anticholinergics (however, local administration is allowed)

    º Cholinergic agents (however, local administration is allowed)

    º Glucocorticosteroids (however, local administration is allowed)

    º Gastrin receptor antagonist, other drugs for the treatment of peptic ulcer

    <Drugs prohibited from Visit 1 to EOT>

    º Rilpivirine, atazanavir, and nelfinavir

    º Antipsychotics, antidepressants, and antianxiety drugs

    <1 week prior to the date of upper gastrointestinal endoscopy(EGD)>

    º Non-steroidal anti-inflammatory drugs (NSAIDs)

    º Antithrombotic agents: Anticoagulants or antiplatelet drugs

    However, among the above drugs, drugs administered as a pre-treatment for upper gastrointestinal endoscopy or for an urea breath test are allowed

    : midazolam, propofol, simethicone, hyoscine butylbromide, cimetropium bromide, magmil, pethidine, gasocol, urea, etc.
16. Subjects who have participated in another clinical trial within 4 weeks from Visit 1 and have been administered with or used an IP or medical device at least once
17. Subjects who have received H.pylori eradication treatment within 4 weeksfrom the date of upper gastrointestinal endoscopy.
18. Subjects who have clinically significant abnormal electrocardiogram

    [Laboratory Tests]
19. Blood test results meet the criteria below at Visit 1:

    º ALT, AST, ALP, GGT, Total bilirubin > 2.0 x ULN

    º eGFR < 60 mL/min/1.73 m2

    [Other]
20. Subjects who cannot undergo upper gastrointestinal endoscopy
21. Pregnant or breast-feeding women
22. Women and men of childbearing potential who are unwilling to use an appropriate medically acceptable method of contraception during the entire study period (Visit 1 through the end of study visit)
23. Subjects who are judged unsuitable for participation in this trial by the investigators for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Cumulative complete healing rate for ulcer confirmed by upper gastrointestinal endoscopy by Week 8 | Week 8

SECONDARY OUTCOMES:
Complete healing rate for ulcers confirmed by upper gastrointestinal endoscopy at Week 4 | Week 4
Complete healing rate for ulcer confirmed by upper gastrointestinal endoscopy at Week 4 by Helicobacter pylori infection status | Week 4
Cumulative complete healing rate for ulcer confirmed by upper gastrointestinal endoscopy according to Helicobacter pylori infection status by Week 8 | Week 8
Changes of Gastrointestinal symptoms per NDI-K at week 4 and 8 | Week 4 and 8
  The frequency and severity of 15 gastointestinal symptoms were scored on a scale from 0 to 4 using a score sheet.
Changes in quality of life (EQ-5D-5L) at Weeks 4 and 8 | Week 4 and 8
Changes and the proportion of changes of the ulcer size(s) at week 4 and week 8 | Week 4 and 8
  Subjects will also rate their health status on the visual analogue scale (VAS) between 0 (the worst state) and 100 (the best state) to get the score for their overall health.
Change of the number of ulcer(s) at week 4 and week 8 | Week 4 and 8

OTHER OUTCOMES:
Exploratory Endpoints | 2weeks after the end of treatment
  Blood Gastrin Test

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Kuro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park KS, Kim HS, Oh JH, Chung WC, Choi SC, Lee SH, Kim TH, Cheung DY, Baik GH, Kim SM, Lee HL, Moon JS, Choi CW, Sohn C, Kim KO, Kim BW, Jung HK, Jung DH, Kim SS, Park MI, Lee JY, Kim GH, Moon HS, Chun H, Shim KN, Shin WG, Park CH, Kim T, Jung SW, Kim H, Jee SR, Lee K, Cho YK, Park SC, Cho J, Huh C, Kwon H, Kim J, Kim J, Park JJ. Randomized, Double-Blind, Active-Controlled, Parallel, Phase 3 Clinical Trial for Evaluating the Efficacy and Safety of Zastaprazan in Patients with Gastric Ulcers. Gut Liver. 2026 Jan 16. doi: 10.5009/gnl250334. Online ahead of print. PMID 41540828